CLINICAL TRIAL: NCT03348280
Title: Vitamin D and Immune Mechanisms of Hypertension in Type 2 Diabetics
Acronym: VDIM
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201707063
Record Dates: First submitted 2017-10-23; First posted 2017-11-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Vitamin D Deficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Vitamin D Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamin D Deficient: Type 2 diabetics with high blood pressure and 25-hydroxyvitamin D levels of <20 ng/ml
  Interventions: Diagnostic Test: Blood draw
- Vitamin D Sufficient: Type 2 diabetics with high blood pressure and 25-hydroxyvitamin D levels of >30 ng/ml
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — Blood will be drawn to isolate monocytes after 2 weeks off of blood pressure lowering medications.

SUMMARY:
This trial will evaluate whether a particular type of circulating white blood cell, monocytes, from type 2 diabetics with high blood pressure and vitamin D deficiency vs. sufficiency will induce hormones that increase blood pressure.

DETAILED DESCRIPTION:
More than half of patients with type 2 diabetes mellitus develop hypertension, which doubles their risk for cardiovascular disease. Inflammation plays a role in the development of these diseases, and monocytes, a type of white blood cell, may be critical. This study will isolate monocytes from blood samples of patients with type 2 diabetes and high blood pressure who have either high levels of vitamin D or low levels of vitamin D, and determine what their effects are on stimulating production in kidney cells of a hormone that increases blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (T2DM)
* Age: 25-80 years old
* Vitamin 25(OH)D3 levels <20 or >30 ng/ml.
* HbA1c: 5.5%-9.5%
* Blood Pressure: <160/100 mm Hg on BP lowering medications and
* Blood Pressure: >120/80 to 160/100 mmHg without BP lowering medications

Exclusion Criteria:

* Recent weight loss of more than 5% within 3 months prior to screening
* Current Pregnancy
* Hypercalcemia
* Previous heart attack and stroke
* Heart failure
* Atrial fibrillation
* Heavy alcohol consumption
* Extreme diets (Atkins, South Beach)
* Chronic renal failure: stage 4 or worse
* >2 + proteinuria on urine sample
* Chronic diseases known to affect immunity

Ages: 25 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: T2DM patients with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Renin production by monocytes | 2 weeks
  Blood will be collected for isolation of monocytes. These cells will then be cultured to determine whether there is monocyte stimulation of a hormone that induces high blood pressure (renin) in kidney cells.

SECONDARY OUTCOMES:
Renin production by monocyte media | 2 weeks
  Blood will be collected for isolation of monocytes. The media from these cells will then be added to culture to determine whether there is stimulation of a hormone that induces high blood pressure (renin) in kidney cells.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Bernal-Mizrachi, MD, Study Director — Washington University School of Medicine
Locations (2):
- United States (2):
  - Barnes-Jewish & Washington University Diabetes Center, St Louis, Missouri
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No